CLINICAL TRIAL: NCT00370903
Title: Retrospective Study of Relationship of Postpartum Depression to Planned Versus Emergent Cesarean Section
Brief Title: Postpartum Depression and Cesarean Section
Status: Completed | Type: Observational
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Other Study IDs: 2005009
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2008-02-04 (Estimated); Status verified 2008-01

CONDITIONS: Postpartum Depression
Keywords: cesarean; planned; emergent; postpartum depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The purpose of this retrospective study is to determine if there is an increase in postpartum depression (PPD) among women who undergo an emergency cesarean section as opposed to a planned cesarean section. We will analyze the hospital and clinic medical records of postpartum women who delivered by cesarean section (CS) at Tulsa Regional Medical Center between January 1, 2003, and June 1, 2005, and who obtained their postpartum care at the OSU Ob/Gyn Clinic in Tulsa, Oklahoma. We will record whether the cesarean was planned or emergent, and we will note the score they received on the Edinburgh Postnatal Depression Scale when they came to the clinic for their four-week postpartum visit. A score of 12 or lower on the EPDS will be considered "not depressed", and a score of 13 or higher will be considered "depressed." Numbers of depressed patients will be compared among the two types of cesarean sections and analyzed for statistical differences using the chi-squared method of analysis.

DETAILED DESCRIPTION:
The purpose of this retrospective study is to determine if there is an increase in postpartum depression (PPD) among women who undergo an emergency cesarean section as opposed to a planned cesarean section. All previous research documenting the rate of PPD in cesarean section patients looks only at the incidence of PPD in cesarean section versus vaginal delivery, and does not separate emergent versus planned cesarean section. The general study hypothesis is as follows: An emergent cesarean section can be an emotionally traumatic experience. Women who have a cesarean section for emergent causes are not psychologically prepared for surgery, and thus experience an increased rate of PPD. The null hypothesis is: There is no significant difference in the rate of PPD among women who have a cesarean section for emergent causes versus women who have their cesarean section at the previously scheduled time.

Postpartum depression (PPD) is diagnosed in approximately 10-20% of women (DSM-IV-TR), and 25% of these women still suffer from PPD twelve months after delivery (Gregoire et al, 1996). Risks for developing PPD include a higher subjective burden of childbirth, poor relationship with spouse, significant other, or father of the baby, unemployment or dissatisfaction with job, and low socioeconomic status.

Obstetrical history risk factors include previous abortions, high-risk pregnancy, low birth weight, and cesarean section (Bergant et al, 1998).

Delivery via cesarean section (CS) creates a much different emotional experience than does a vaginal delivery. Disappointment in the ability to have a natural birth, feelings of resentment towards the physician, altered treatment expectation, as well as, pain and trauma associated with surgery are all contributing factors (Al-Nuaim, 2004). A majority of women consider an emergency cesarean section (CS) to be a mentally traumatic encounter. One third of women who require an emergency CS will experience posttraumatic stress reactions during the postpartum period (Ryding et al, 1997). Fisher et al reported that there is a significant relationship between mode of delivery and negative psychological outcomes. A mother who has a CS instead of a vaginal delivery is more likely to have mood deterioration, lowered self-esteem, grief reaction, posttraumatic distress, and depression (Fisher et al, 1997).

We propose to analyze the hospital and clinic medical records of 200 postpartum women who delivered by cesarean section (CS) at Tulsa Regional Medical Center between January 1, 2003, and June 1, 2005, and who obtained their postpartum care at the OSU Ob/Gyn Clinic in Tulsa, Oklahoma. Of the charts reviewed, 100 women will have had a CS for emergent causes, and the other 100 will have delivered via a planned CS.

The hospital records will be reviewed to determine whether the cesarean delivery was for emergent causes or if it was a planned operation. Planned cesarean sections are performed on patients who have had a previous CS and are scheduled for a repeat, fetuses that are measuring greater than 4000 grams, prior uterine scars, and known breech presentations on patients not in labor. Emergent causes will include nonreassuring fetal heart tones, placental abruption, inductions that result in CS due to failure to progress or cephalopelvic disproportion, and malpresentations in active labor. Malpresentations include face, brow, shoulder, hand, breech, compound, or transverse lie.

The patients will have their clinic chart reviewed for the following data from their antenatal and postpartum visits: date of delivery, breastfeeding status as a simple yes/no question without regard to whether or not the mother is supplementing with formula, mother's age, smoker/non-smoker, race, employment status, previous history psychological disorders, Edinburgh Postnatal Depression Scale score (routinely administered by obstetrician at the six week postpartum visit), other antepartum or postpartum complications.

Postpartum depression will be diagnosed with the assistance of the Edinburgh Postnatal Depression Scale (EPDS). The OSU Ob/Gyn Clinic began routine use of the EPDS in 2003. As a result, all patient records used in this study will be from January 1, 2003 to June 1, 2005. A one-year time period has been allotted for collection of data as this will allow sufficient time to review the necessary records. In addition, one of the collaborating investigators is a resident, and the research assistants are medical students, therefore, the data collection must be completed in a timely manner. OSU Ob/Gyn and Tulsa Regional Medical Center are the only sites in this investigation to ensure that the diagnosis of postpartum depression is made using the same parameters.

STUDY POPULATION

Inclusion/Exclusion Criteria

Our study population will include 200 postpartum women ages 15 to 43 who have given birth via cesarean section at Tulsa Regional Medical Center. In addition, these same individuals must have had their postpartum follow up visit(s) at the OSU Ob/Gyn Clinic in Tulsa, Oklahoma. The study population consists predominantly of Medicaid patients. These patients are generally of a lower socioeconomic status. The ethnic mix includes Caucasian, African-American, Hispanic, American Indian and Asian patients. Patients who deliver vaginally, have an intrauterine fetal demise, known anomalies in the delivered fetus, a known mood disorder during pregnancy, or drug use during pregnancy or the postpartum course will be excluded.

Early Termination Criteria

N/A

METHODS/PROCEDURES

Diagnosis

The diagnosis of postpartum depression will be given based on the use of the Edinburgh Postnatal Depression Scale (EPDS). The EPDS has 10 questions, and possible scores range from 0-30. We used its author's recommendation that scores higher than 12 be considered a positive screen for PPD and for which sensitivity and specificity have been found to be 86% and 78%, respectively (Cox et al). We are aware that other depression evaluations may be used to definitively diagnose PPD. The OSU Ob/Gyn clinic uses the EPDS for convenience, and it was the only data available in patient charts for this retrospective study.

DATA

Collection Collaborating investigators and research assistants will review each chart, and extract only the following data from the patient's postpartum visit: Edinburgh Postnatal Depression Scale score (routinely administered by obstetrician at the six week postpartum visit), breastfeeding status as a simple yes/no question without regard to whether or not the mother is supplementing with formula, date of delivery, mother's age, smoker/non-smoker, race, employment status, previous history psychological disorders, other antepartum or postpartum complications. No additional information will be collected from patient charts. The research assistants are OSU medical students employed in the work study program for the specific purpose of working on this research project. They will collect the data from clinic records. These assistants are under the OSU umbrella of individuals who may have access to patient charts, and they have basic human use research training as well as HIPAA training.

Analysis Numbers of depressed patients will be compared among the two groups and analyzed for statistical differences using the chi-squared method of analysis.

Confidentiality Patient's clinic records will be kept in the medical records department, which is under direct security supervision, or locked at all times. Hospital records will be kept in the health information management department at Tulsa Regional Medical Center, which is locked 24 hours a day. All study records will be de-identified by conversion to numbers before review, analysis, or interpretation. J. Martin Beal, D.O., Sarah McCoy, Ph.D., and Jennifer Howell, D.O. will have access to these numbers which will be kept locked in the OSU Ob/Gyn office, which is separate from both medical records departments. All documents linking patient names to charts will be destroyed after the data collection is complete.

ELIGIBILITY:
Inclusion Criteria:

* Included are postpartum women ages 15 to 43 who have given birth via cesarean section at Tulsa Regional Medical Center between January 1, 2003 and June 1, 2005. Postpartum follow up visit(s) must have occurred at the OSU Ob/Gyn Clinic in Tulsa, Oklahoma.

Exclusion Criteria:

* Patients who deliver vaginally, have an intrauterine fetal demise, known anomalies in the delivered fetus, a known mood disorder during pregnancy, or drug use during pregnancy or the postpartum course will be excluded.

Ages: 15 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200
Dates: Start 2006-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M. Beal, D.O., Principal Investigator — Oklahoma State University Center for Health Sciences
Locations (1):
- Oklahoma State University Center for Health Sciences Houston Parke Clinic, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] Ryding EL, Wijma B, Wijma K. Posttraumatic stress reactions after emergency cesarean section. Acta Obstet Gynecol Scand. 1997 Oct;76(9):856-61. doi: 10.3109/00016349709024365. PMID 9351412